CLINICAL TRIAL: NCT05546905
Title: An Observational Study Describing Diagnosis and Treatment Patterns in Adults With Metastatic Non-small Cell Lung Cancer With BRAF V600E Mutation in Clinical Practice, to Assess Treatment Effectiveness and Quality of Life (OCTOPUS)
Brief Title: A Study in Patients With BRAF V600E-mutant Metastatic Non-small Cell Lung Cancer (OCTOPUS)
Status: Completed | Type: Observational
Sponsor: Pierre Fabre Medicament (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS12500
Record Dates: First submitted 2022-06-23; First posted 2022-09-21 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Non-small Cell Lung Cancer; BRAF V600 Mutation
Keywords: Metastatic Non-small Cell Lung Cancer; BRAF V600 Mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to describe the treatment patterns in clinical practice in adult patients with mNSCLC with a BRAF V600E mutation. This study will also describe Real-World Progression-Free Survival (rwPFS) and Overall Survival (OS) for treatments prescribed in routine practice for mNSCLC with BRAF V600E mutation. Adverse events (AEs) related to treatment management will also be described.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of first-line treatment initiation for mNSCLC,
* Patients who initiated a first systemic treatment for mNSCLC in the metastatic setting from 01 December 2017 and before their study entry date (retrospectively enrolled patients), or Patients who initiated a first systemic treatment for mNSCLC (metastatic setting) at or after their study entry date (prospectively enrolled patients),
* Confirmed diagnosis of Stage IV mNSCLCat any time before study inclusion Stage IV M1a, M1borM1c, as per the American Joint Committee on Cancer (AJCC cancer) staging manual,
* Confirmed presence of BRAF V600E mutation - via tumor biopsy, metastasectomy, or liquid biopsy - at anytime before study inclusion,
* Signed ICF or non-opposition to study participation,according to local regulations.

Patients eligible for prospective QoL data collection must, in addition to the above mentioned criteria, meet ALL of the following criteria to be eligible for the study:

* Patients who initiate a first or second systemic treatment line for mNSCLC (metastatic setting) with a BRAF V600E mutation at or after their study entry date

Exclusion Criteria:

* Concurrent or another previous malignancy within 2 years of study entry, except curatively treated basal or squamous cell skin cancer, prostate intraepithelial neoplasm, in-situcarcinoma of the cervix, Bowen's disease or Gleason ≤ 6 prostate cancer,
* Previous, ongoing, or planned participation in a clinical trial involving an interventional drug as a first-or second-line systemic treatment for mNSCLC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients diagnosed with mNSCLC BRAF V600E mutation who initiated a 1st systemic (retrospectively enrolled patients), and patients who initiated a first metastatic treatment upon inclusion (prospectively enrolled patients). Retrospectively enrolled patients can also be eligible for second-line prospective QoL data collection and contribute to a sub-cohort of prospective patients initiating their 2nd line of treatment (LoT) after study entry. The study aims to enroll approximately 200 patients, of whom 50 patients are planned to complete full prospective follow-up for their first-line and/or second-line systemic treatment given in the metastatic setting in mNSCLC allowing for prospective QoL data collection.
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Description of treatment regiment/agents for first and second systemic treatment lines for mNSCLC | From the start of first or second line treatment to progression or date of death from any cause,assessed up to 30 months
  Names of regimens/agents
Description of line of treatment | From the start of first or second line treatment to the end of second line treatment,assessed up to 30 months
  Line of treatment number overall, not limited to metastatic setting
Description of duration of treatment line | From the start of first or second line treatment to the end of line treatment,assessed up to 30 months
  Duration of treatment line = End date of treatment line - Start date of treatment line
Time to treatment discontinuation | From the start of first or second line treatment to the treatment discontinuation or death,assessed up to 30 months
  Time to treatment discontinuation defined as the time between the date of start of a medication and the date of treatment discontinuation or death.
Time to next treatment | From the start of first or second line treatment to the subsequent line treatment,assessed up to 30 months
  Time to next treatment defined as the time between the date of start of a medication and the date of start of the next LoT.

CONTACTS AND LOCATIONS:
Overall Officials: François Denjean, Study Director — Pierre Fabre Médicament
Locations (39):
- France (9):
  - CHU Lyon - Hôpital Cardio-Vasculaire et Pneumologique Louis Pradel, Lyon, Auvergne-Rhône-Alpes
  - CHU Angers - Hôpital Larrey, Angers
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre Hospitalier de Douai, Douai
  - CHU Nantes - Hôpital Guillaume et René Laënnec, Nantes
  - CHU Poitiers - Hôpital la Milétrie, Poitiers
  - CHU Rennes - Hopital Pontchaillou, Rennes
  - CHU Strasbourg - Nouvel Hôpital Civil, Strasbourg
  - UNEOS - Hopital Robert Schuman, Vantoux
- Germany (6):
  - Kliniken Essen-Mitte, Essen
  - Universitaetsklinikum Giessen und Marburg GmbH Standort Giessen, Giessen
  - Marienhaus Klinikum Mainz, Mainz
  - Kliniken Maria Hilf GmbH, Mönchengladbach
  - LMU-Campus Innenstadt, München
  - Thoraxzentrum Unterfranken, Münnerstadt
- Italy (10):
  - Azienda Ospedaliera Nazionale Santi Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda Ospedaliera San Giuseppe Moscati, Avellino
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII (Presidio Papa Giovanni XXIII), Bergamo
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Presidio Spedali Civili), Brescia
  - IRCCS Istituto Scientifico Romagnolo Per Lo Studio e La Cura Dei Tumori "Dino Amadori" - IRST, Meldola
  - Azienda Socio Sanitaria Territoriale Niguarda (Grande Ospedale Metropolitano Niguarda), Milan
  - AOU Cagliari- P.O. Policlinico Universitario Duilio Casula, Monserrato
  - Azienda Ospedaliera Universitaria- Università degli Studi della Campania "Luigi Vanvitelli", Napoli
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
- Spain (11):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - ICO Badalona - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Universitario HM Madrid Sanchinarro, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
  - Fundacion Hospital Son Llatzer, Palma de Mallorca
  - Complejo Hospitalario Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
- United Kingdom (3):
  - Royal Marsden Hospital- London, London
  - Nottingham University Hospitals City Campus, Nottingham
  - Velindre Cancer Centre, Whitchurch